CLINICAL TRIAL: NCT06411080
Title: UltraSound Evaluation of Fluid tOleRanCE for Acute Kidney Injury: A Pilot Randomized Controlled Trial
Brief Title: UltraSound Evaluation of Fluid tOleRanCE for Acute Kidney Injury
Acronym: USE-the-FORCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2025-12250
Record Dates: First submitted 2024-05-08; First posted 2024-05-13 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-09

CONDITIONS: Acute Kidney Injury
Keywords: point-of-care ultrasound; VExUS; Lung ultrasound; Fluid therapy; acute kidney injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Management with ultrasound information (Experimental): An ultrasound report will be provided to the attending care team. The report will contain information related to abdominal and thoracic ultrasound exams with expert interpretation regarding anticipated risks of fluid administration.
  Interventions: Diagnostic Test: Ultrasound evaluation of fluid tolerance
- Usual care (No Intervention): Usual care without information from Point-Of-Care ultrasound assessment of fluid tolerance.

INTERVENTIONS:
Diagnostic Test: Ultrasound evaluation of fluid tolerance — Lung ultrasound for the assessment of B-line artifact and pleural effusion combined with abdominal ultrasound for VExUS assessment. The imaging study will be reviewed by an expert for will generate a report with interpretation regarding the risk of fluid administration. The assessment will be performed at baseline and after 48 hours after randomization.
  Arms: Management with ultrasound information

SUMMARY:
Fluid expansion with isotonic crystalloids is a first-line intervention in the treatment of patients with acute kidney injury (AKI). While it is generally accepted that the timely correction of kidney hypoperfusion will minimize the extent of injury as well as potentially facilitate recovery, there are potential harms involved in indiscriminate administration of intravenous fluids. Although anticipating fluid tolerance is part of the clinical evaluation of a patient for whom intravenous fluid therapy is considered, it has been suggested that using Point-Of-Care ultrasound (POCUS) may enable the early identification of patients with a high-risk of congestive complications and guide clinical decisions with greater precision[1]. However, it has not been shown that providing this information in the context of AKI result in a change in management or a prevention of complications.

This single-center pilot randomized controlled trial aim to determine the feasibility of comparing a management including a POCUS evaluation of fluid tolerance to usual care in non-critically ill patients with AKI. In the intervention group, a POCUS evaluation will be performed and interpreted by experienced staff producing a report that will be presented to the attending care team. This assessment will be repeated 48-72 hours later. The primary aim of the study will be to establish the feasibility of this intervention. Secondary objectives will include determining the difference between the intervention arm and the control arm in relationship with fluid administration, diuretic use, evolution of kidney function, and intensification of care.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ 18 year-old
2. Admitted to the hospital
3. Acute kidney injury defined by the KDIGO criteria[48]
4. Fluid expansion is considered by attending nephrologist or already ongoing

Exclusion Criteria:

1. Admitted to the intensive care unit
2. Known stage 5 chronic kidney disease according to the KDIGO classification receiving renal replacement therapy or not.
3. Renal replacement therapy for AKI has been initiated or is planned within 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-10-17 (Actual); Primary Completion 2025-09-29 (Actual); Study Completion 2025-10-22 (Actual)

PRIMARY OUTCOMES:
Protocol adherence | 30 days
  : Ultrasound assessments were performed as planned and the reports were generated and transmitted to the attending care team in the prespecified periods.

SECONDARY OUTCOMES:
Cumulative intravenous fluid | 5 days
  Amount of fluid in mL received
Diuretic use | 5 days
  defined as the use of loop diuretics
Kinetic estimated glomerular filtration rate (KeGFR) | 5 days
  Kinetic estimated glomerular filtration rate (KeGFR) will be derived from serial measurements in serum creatinine
Progression to a higher stage of AKI | 5 days
  Progression to a higher stage of AKI will be defined as any increase in the KDIGO staging criteria of increase in creatinine:
  Operational definition: Increase in at least one level compared to baseline AKI staging during the first 5 days:
  Stage 1: Increase in serum creatinine by ≥26.5 µmol/L within 48 hours or increase to 1.5-1.9 times baseline within the last 7 days.
  Stage 2: Increase in serum creatinine to 2.0-2.9 times baseline. Stage 3: Increase in serum creatinine to ≥3.0 times baseline or increase to ≥354 µmol/L, Stage 3D: Initiation of renal replacement therapy.
Death or escalation of care | 10 days
  composite endpoint defined as the occurrence of at least one of the following events occurring within 10 days after randomization: death from any cause, intervention of the rapid response team, admission to the intensive care unit, initiation of non-invasive positive pressure ventilation, initiation of renal replacement therapy. (Binary - Yes/no)

OTHER OUTCOMES:
Kidney and liver stiffness | 5 days
  median values of shear-wave propagation speed in m/sec obtained by shear-wave elastography assessment of the respective organ parenchyma.
The perceived usefulness of the ultrasound report | 5 days
  be reported on a sliding scale from 0 to 5. A score of 0 will mean that the information is considered useless while a score of 5 will mean that the information provided had a critical impact of clinical management. (Continuous - points)

CONTACTS AND LOCATIONS:
Overall Officials: William Beaubien-Souligny, MD PhD, Principal Investigator — Centre Hospitalier d'Université de Montréal
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No